CLINICAL TRIAL: NCT06736223
Title: A Multicentric, Open-label, Non-randomized Study to Evaluate the Pharmacokinetic, Safety and Tolerability of ITF2357 Given as an Oral Single 50 mg Dose in Participants With Chronic Hepatic Impairment Relative to Matched Participants With Normal Hepatic Function
Brief Title: Pharmacokinetics, Safety and Tolerability of ITF2357 in Participants With Chronic Hepatic Impairment and With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ITF/2357/60; 2024-513577-43-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment
MeSH Terms: interventions — givinostat hydrochloride; givinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild HI (Experimental): Patients with mild HI (Child-Pugh class A)
  Interventions: Drug: ITF2357
- Moderate HI (Experimental): Patients with moderate HI (Child-Pugh class B)
  Interventions: Drug: ITF2357
- Healthy Volunteers (Experimental): Participants with normal hepatic function (control group)
  Interventions: Drug: ITF2357

INTERVENTIONS:
Drug: ITF2357 — ITF2357 (INNM Givinostat hydrochloride Monohydrate), single dose
  Other Names: Givinostat; Givinostat hydrochloride Monohydrate

SUMMARY:
This is a multicentric, open-label, non-randomized study to evaluate the pharmacokinetic, safety and tolerability of ITF2357 in participants with chronic hepatic impairment relative to matched participants with normal hepatic function.

DETAILED DESCRIPTION:
This study will evaluate the effect of mild and moderate hepatic impairment (HI) on the pharmacokinetics of ITF2357 and its metabolites.

The total number of participants to be enrolled in the study is 24 subjects:

* 8 Participants with mild HI (Child-Pugh class A)
* 8 Participants with moderate HI (Child-Pugh class B)
* 8 Participants with normal hepatic function (control group)

Each participant will go through:

* A screening period from Day (D)-28 to D-2
* One 6-day/5-night inpatient period (from D-1 evening to D5 morning)
* An end-of-study evaluation to be done on D10 (±1 day).

ELIGIBILITY:
Inclusion Criteria for Participants with HI:

1. Male or female participants, between 18 and 75 years of age, inclusive.
2. Body weight between 60.0 and 110.0 kg, inclusive if male, and between 50.0 and 100.0 kg, inclusive if female, body mass index (BMI) between 18.00 and 34.99 kg/m2, inclusive.
3. Stable chronic liver disease assessed by medical history, physical examination, laboratory values.
4. Vital signs after 10 minutes resting in supine position within the following range [or if out of range, considered not clinically significant (NCS) by the Investigator]:

95 mmHg < systolic blood pressure (SBP) < 180 mmHg 45 mmHg < diastolic blood pressure (DBP) < 100 mmHg 40 bpm < heart rate (HR) < 100 bpm. 5. 12-lead ECG without clinically significant abnormality, in the judgment of the Investigator; in no circumstances should participants be enrolled with corrected QT according to Fridericia (QTcF) > 450 ms.

6. Laboratory parameters within the acceptable range for participants with HI; however, serum creatinine should be strictly below the upper laboratory range.

7. Female participants who are not pregnant or nursing at Screening and Day -1, or who are not planning to become pregnant during study period and until 4 weeks after the IMP administration.

8. Female participants of non-childbearing potential, defined as one of the following:

a. At least 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., appropriate age) and follicle-stimulating hormone (FSH) in the range for menopausal female confirmed by blood test according to current local standards at screening.

b. Those with history of hysterectomy or surgical removal of both ovaries or bilateral tubal ligation performed at least 90 days prior to Screening.

9. Female participant of childbearing potential and male participant must agree to use an adequate and highly effective method of contraception (according to Clinical Trials Coordination Group [CTCG] recommendations) during the study and for at least 90 days after the study drug administration for women and for men. Such methods include:

1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation oral, intravaginal or transdermal.
2. progestogen-only hormonal contraception associated with inhibition of ovulation oral, injectable or implantable
3. intrauterine device (IUD)
4. intrauterine hormone-releasing system (IUS)
5. bilateral tubal occlusion
6. vasectomized partner
7. sexual abstinence (when in line with the preferred and usual subject's lifestyle).

   Note: Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM) are not acceptable methods of contraception.

   10. Having given written informed consent prior to any procedure related to the study.

   11. Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.

   12. Not under any administrative or legal supervision. 13. For moderate HI cohort: Child-Pugh total score ranging from 7 to 9, inclusive.

   14. For mild HI cohort: Child-Pugh total score ranging from 5 to 6, inclusive. 15. Male participants must agree not to donate sperm from inclusion up to 3 months after ITF2357 dosing.

   Exclusion Criteria for Participants with HI:
   1. Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecological (if female), or infectious disease, or signs of acute illness.
   2. Hepatocarcinoma.
   3. Acute hepatitis.
   4. Hepatic encephalopathy grade 2, 3, and 4.
   5. Blood donation within 2 months before inclusion.
   6. Symptomatic postural hypotension, whatever the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in SBP ≥ 30 mmHg within 3 minutes when changing from supine to standing position.
   7. Presence or history of drug hypersensitivity, or allergic disease, except seasonal rhinitis, diagnosed and treated by a physician.
   8. History or presence of regular use of recreational drugs or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis) within 2 years before inclusion.
   9. Smoking more than 15 cigarettes or equivalent per day, unable to refrain from smoking over 5 cigarettes per day from D-1 and throughout the entire institutionalization (i.e., up to D5).
   10. Excessive consumption of beverages with xanthine bases (more than 4 cups or glasses per day).
   11. If female, pregnancy [defined as positive β-human choriogonadotropin (β-HCG) blood test] or breast feeding.
   12. Any significant change in chronic treatment medication within 14 days before inclusion.
   13. Consumption of PgP or BCRP potent inducers or inhibitors that could impact the PK of the investigational product.
   14. Any vaccination, including COVID-19 within 2 weeks before inclusion.
   15. Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
   16. Any participant in the exclusion period of a previous study according to applicable regulations.
   17. Any participant who cannot be contacted.
   18. Any participant who is the Investigator or any co-Investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
   19. Positive result on any of the following tests: anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
   20. Positive results on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates) unless this result is secondary to a documented medical prescription (only for benzodiazepines and cannabinoids).
   21. Positive alcohol breath test.
   22. Any consumption of citrus fruits (grapefruit, Seville orange, etc.) or their juices within 5 days before inclusion.
   23. Medications that prolong the QTc Interval (refer to the list provided in the Appendix 12) within 14 days before inclusion or within 7 times the elimination half-life before inclusion.

   Note: If any of those drugs is planned to be administered in any of the potential participants, it needs to be postponed for at least until the last ECG at EOS is completed.

   Inclusion Criteria for Participants with normal hepatic function:
   1. Male or female participants, between 18 and 75 years of age, inclusive.
   2. Body weight within 10% of the mean body weight of the participants with HI to be matched, and BMI between 18.00 and 34.99 kg/m2, inclusive.
   3. Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
   4. Vital signs after 10 minutes resting in the supine position within the following range (or if out of range, considered NCS by the Investigator):

   95 mmHg < SBP < 140 mmHg 45 mmHg < DBP < 90 mmHg 40 bpm < HR < 100 bpm. 5. 12-lead ECG without clinically significant abnormality, in the judgment of the Investigator; in no circumstances should participants be enrolled with QTcF > 450 ms.

   6. Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy participants, except in the case of platelets, white blood cells and hemoglobin below lower limit of normal (LLN); however serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the participant has documented Gilbert's syndrome, with a maximum bilirubin level lower than 3 x [upper limit of normal (ULN)] and any parameter for which there is an explicit stopping rule should not exceed the upper laboratory range.

   7. Female participants who are not pregnant or nursing at Screening and Day -1, or who are not planning to become pregnant during study period and until 4 weeks after the IMP administration.

   8. Female participants of non-childbearing potential, defined as one of the following:

a. At least 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., appropriate age) and follicle-stimulating hormone (FSH) in the range for menopausal female confirmed by blood test according to current local standards at screening.

b. Those with history of hysterectomy or surgical removal of both ovaries or bilateral tubal ligation performed at least 90 days prior to Screening.

9. Female participant of childbearing potential and male participant must agree to use an adequate and highly effective method of contraception (according to CTCG recommendations) during the study and for at least 90 days after the study drug administration for women and for men. Such methods include:

1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation oral, intravaginal or transdermal.
2. progestogen-only hormonal contraception associated with inhibition of ovulation oral, injectable or implantable
3. intrauterine device (IUD)
4. intrauterine hormone-releasing system (IUS)
5. bilateral tubal occlusion
6. vasectomized partner
7. sexual abstinence (when in line with the preferred and usual subject's lifestyle).

   Note: Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and LAM are not acceptable methods of contraception.

   10. Having given written informed consent prior to any procedure related to the study.

   11. Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.

   12. Not under any administrative or legal supervision. 13. Male participants must agree not to donate sperm from inclusion up to 3 months after ITF2357 dosing.

   Exclusion Criteria for Participants with HI:
   1. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecological (if female), or infectious disease, or signs of acute illness.
   2. Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
   3. Blood donation within 2 months before inclusion.
   4. Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in SBP ≥ 20 mmHg within 3 minutes when changing from supine to standing position.
   5. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician, except seasonal rhinitis.
   6. History or presence of regular use of recreational drugs or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis) within 2 years before inclusion.
   7. Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking from D-1 and throughout the entire institutionalization (i.e., up to D5).
   8. Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
   9. If female, pregnancy (defined as positive β-HCG blood test), breast-feeding.
   10. Any medication (including PgP or BCRP inducers or inhibitors, or omeprazole) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic (PD) half-life of the medication (except HRT and contraception when applicable), any vaccination within the last 28 days (except COVID-19 vaccination) and any biologics (antibody or its derivatives) given within 4 months before inclusion.
   11. Any vaccination, including COVID-19 within 2 weeks before inclusion.
   12. Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
   13. Any participant in the exclusion period of a previous study according to applicable regulations.
   14. Any participant who cannot be contacted.
   15. Any participant who is the Investigator or any co-Investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
   16. Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-HIV1 and anti HIV2 Ab.
   17. Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
   18. Positive alcohol breath test.
   19. Any consumption of citrus (grapefruit, Seville orange, etc.) or their juices within 5 days before inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration observed (Cmax) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Area under the plasma concentration versus time curve to the real time tlast (AUClast) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Area under the plasma concentration versus time curve extrapolated to infinity (AUC0-inf) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose

SECONDARY OUTCOMES:
Time to reach Cmax (tmax) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Apparent terminal half-life (t1/2) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Apparent total plasma clearance from plasma (CL/F) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Apparent volume of distribution (Vz/F) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Maximum plasma concentration observed (Cmax) of ITF2357 metabolites | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Area under the plasma concentration versus time curve to the real time tlast (AUClast) of ITF2357 metabolites | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Area under the plasma concentration versus time curve extrapolated to infinity (AUC0-inf) of ITF2357 metabolites | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Time to reach Cmax (tmax) of ITF2357 metabolites | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Apparent terminal half-life (t1/2) of ITF2357 metabolites | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Unbound fraction (fu) of ITF2357 and its metabolites | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Unbound area under the plasma concentration time curve (AUCu) of ITF2357 and its metabolites | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Unbound maximum plasma concentration observed (Cmax,u) of ITF2357 and its metabolites | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Unbound apparent total plasma clearance (CL/Fu) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Unbound apparent volume of distribution (Vz/Fu) of ITF2357 | Pre-dose (30 minutes before administration), then 0.5 to 96-hour post-dose
Electrocardiogram QT interval corrected according to Fredericia's formula (ECG QTcF) | From Baseline (28 to 2 days before administration) to End of Study (9 to 11 days after administration)
Incidence of Treatment Emergent Adverse Events (TEAEs) | From Baseline (28 to 2 days before administration) to End of Study (9 to 11 days after administration)
  Treatment Emergent Adverse Event is defined as any untoward medical occurrence (including an abnormal laboratory finding, symptom or a disease) in a participant administered the pharmaceutical product and that does not necessarily have to have a causal relationship with this treatment
Severity of Treatment Emergent Adverse Events (TEAEs) | From Baseline (28 to 2 days before administration) to End of Study (9 to 11 days after administration)
  Treatment Emergent Adverse Event is defined as any untoward medical occurrence (including an abnormal laboratory finding, symptom or a disease) in a participant administered the pharmaceutical product and that does not necessarily have to have a causal relationship with this treatment

CONTACTS AND LOCATIONS:
Locations (2):
- MC COMAC Medical Ltd, Sofia, Bulgaria
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: No